CLINICAL TRIAL: NCT01060384
Title: Phase I/II Study of Lenalidomide and Ofatumumab for the Treatment of Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Study of Lenalidomide and Ofatumumab for the Treatment of Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Celgene Corporation (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0514-09-FB
Record Dates: First submitted 2010-01-25; First posted 2010-02-02 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Lenalidomide; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase 1/Phase II (Experimental): All participants will receive the same dose of Ofatumumab. There will be three planned dose cohorts for the Lenalidomide in the Phase 1 portion of this trial. A maximum of 18 patients will be enrolled in to Phase 1. Three evaluable patients will be enrolled in to each of the dose cohorts with an additional 3 patients to be enrolled in the maximum tolerated dose (MTD). An additional 29 evaluable patients will be enrolled in to Phase II using the MTD for Lenalidomide that was determined in Phase 1.
  Interventions: Drug: Lenalidomide; Drug: ofatumumab

INTERVENTIONS:
Drug: Lenalidomide — Dose Cohort -1^ 10mg daily on Days 1-21 every 28 days
  Dose Cohort +1^^ 15mg daily on Days 1-21, every 28 days
  Dose Cohort +2 20 mg daily on Days 1-21, every 28 days
  Dose Cohort #3 25 mg daily on Days 1-21, every 28 days
  ^Used only if Dose Cohort +1 requires further reduction
  ^^Starting Dose Cohort in Phase I
  Other Names: REVLIMID
Drug: ofatumumab — 8 weekly infusions of ofatumumab 1000mg.
  Other Names: Kesimpta

SUMMARY:
The purpose of this trial is to investigate the efficacy (how well the drug works) of ofatumumab and lenalidomide in patients with lymphoma and to investigate if any possible unwanted side effects may occur. The purpose of the Phase I portion of this trial will be to determine the maximum dose of these medications that can be given with minimal side effects.

DETAILED DESCRIPTION:
This trial will investigate the efficacy of ofatumumab and lenalidomide in patients with lymphoma and investigate if any possible unwanted side effects may occur. Ofatumumab is a human antibody (a type of protein) that binds specifically to a protein (CD20) on the surface of some of the white blood cells (B-cells). Research, so far, has shown that ofatumumab can destroy cancer cells which originate from B cells. Ofatumumab is approved for sale by the US Food and Drug Administration (FDA). The medicine has an approved indication for Chronic Lymphocytic Leukemia (CLL) but is not approved for Non-Hodgkin's Lymphoma (NHL).

Lenalidomide is a drug that affects the immune system. Lenalidomide can change the body's immune system and it may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, it may reduce or prevent the growth of cancer cells. Lenalidomide is approved by the FDA for treatment of multiple myeloma (MM) and myelodysplastic syndrome (MDS) and has been shown to be effective in lymphoma that does not respond to treatment or has come back after treatment. Lenalidomide has not been approved by the United States (US) Food and Drug Administration (FDA) and is experimental (investigational) in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of CD20+ non-Hodgkin's lymphoma that is recurrent or refractory after at least one prior therapy and for which no other potentially curative therapy is available.
* Subject, age > or = 19 years
* Patients must have relapsed or refractory disease after at least one prior systemic therapy, with at least a 3 week interval from the completion of the most recent chemotherapy or radiotherapy regimen (unless the patient has had progressive disease prior to the 3 weeks). Patient has resolved all toxicities to ≤ grade 1, felt to be related to prior therapy.
* Patients must be ineligible or relapsed after an autologous or allogeneic stem cell transplant if clinically appropriate.
* Adequate Laboratory Parameters:

  * ANC ≥ 1500/μL
  * Platelet count ≥75,000/μL
  * Total bilirubin ≤ 1.5 times the institutional Upper Limit of Normal (ULN)- unless due to NHL
  * Hepatic enzymes (AST, ALT ) ≤ 2.5 times the institutional ULN - unless due to NHL
  * Serum Creatinine < 3.0 times the institutional ULN - unless due to NHL
  * Creatinine clearance ≥60ml/min during phase I (See Appendix A) Creatinine clearance ≥ 30ml/min during phase II and patients with creatinine clearance ≥ 30ml/min and < 60ml/min should start Lenalidomide at a reduced dose. See Section 5.3.1
* Females of child-bearing potential (FCBP) must agree to:

Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. See Appendix B: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.

Note: A FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (i.e., amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Male patients must:

* Agree to use a condom during sexual contact with a FCBP, even if they have had a vasectomy, throughout study drug therapy, during any dose interruption and 28 days after cessation of study therapy.
* Agree to not donate semen during study drug therapy and for a period after end of study drug therapy
* ECOG Performance status of 0-2 (See Appendix C)
* Signed written informed consent including HIPAA according to institutional guidelines

Exclusion Criteria:

* No malignancy [other than the one treated in this study] which required systemic treatment within the past 3 years.
* Patients not willing to take DVT prophylaxis
* Pregnant or lactating females
* Positive serology for hepatitis B (HB) defined as positive test of HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded. Patients with documented vaccination against Hepatitis B will not be considered positive.
* Known seropositive for active viral infection with human immunodeficiency virus (HIV), or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Patients with ≥ Grade 2 neuropathy
* Active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Known CNS involvement with lymphoma
* Significant concurrent, uncontrolled medical condition, that in the judgment of the investigator, may affect the patient's ability to sign the informed consent and comply with study procedures.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-03-29 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Saint Francis Medical Center, Grand Island, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the patients will receive 8 weekly infusions of Ofatumumab 1000mg. Dose escalation of Lenalidomide planned in three dose cohorts. Dose reduction Cohort (-1) will be added if severe adverse events noted in 2/3 patients. Phase II will evaluate Lenalidomide at maximum tolerated dose (MTD) and Ofatumumab in 36 patients.
Groups:
- Phase 1: Cohort -1: Cohort -1 received 10 mg Lenalidomide per day on days 1-21 every 28 days.
- Phase 1: Cohort #1: Cohort 1 received 15 mg Lenalidomide per day on days 1-21 every 28 days.
- Phase 1: Cohort #2: Cohort 2 received 20 mg Lenalidomide on days 1-21 every 28 days.
- Phase 1: Cohort #3: Cohort 3 received 25 mg Lenalidomide per day on days 1-21 every 28 days.
- Phase II: Event Free Survival and Overall Survival: Event free and overall survival probabilities will be computed on all patients receiving the MTD dose, including those patients in the phase I portion of the study.
Period: Overall Study
Arm/Group | Phase 1: Cohort -1 | Phase 1: Cohort #1 | Phase 1: Cohort #2 | Phase 1: Cohort #3 | Phase II: Event Free Survival and Overall Survival
Started | 6 | 4 | 0 | 0 | 36
Completed | 6 | 3 | 0 | 0 | 34
Not Completed | 0 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Intercurrent illness | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 1/Phase II: There will be three planned dose cohorts for the Lenalidomide in the Phase 1 portion of this trial. Three evaluable patients will be enrolled in to each of the dose cohorts with an additional 3 patients to be enrolled in the maximum tolerated dose (MTD). Patients will be enrolled in to Phase II using the MTD for Lenalidomide that was determined in Phase 1.
  Dose Cohort -1: 10 mg per day. This cohort will be used only if needed due to dose reduction in Dose cohort +1.
  Dose Cohort +1: 15 mg per day. Dose Cohort +2: 20 mg per day. Dose Cohort +3: 25 mg per day.
  Phase II: An additional 29 response-evaluable patients will be enrolled into Phase II using the MTD for Lenalidomide that was determined in Phase 1.
  All subjects will receive the same dosing schedule for Ofatumumab regardless of which Phase of the trial they are enrolled.
Arm/Group | Phase 1/Phase II
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 63.4 [35.5 to 80.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Lenalidomide
Description: The maximum tolerated dose (MTD) will be defined as the next lowest dose cohort below where ≥ 2/3 or ≥ 3/6 patients experience dose limiting toxicities in cycle 1.
Time Frame: 7 months
Population: Ten patients were enrolled in Phase 1. One patient was inevaluable, thus 9 patients are evaluable for outcome. Patients will be evaluable for Dose Limiting Toxicity (DLT) if they receive at least 75% of the planned doses of study drugs or they experience DLT in cycle 1 or and have sufficient followup data to determine whether DLT occurred.
Measure: Number; unit: milligrams
Groups:
- Phase 1: Maximum Tolerated Dose (MTD) of Lenalidomide
Arm/Group | Phase 1
Number analyzed (Participants) | 9
milligrams | 10

2. Secondary Outcome: Phase I and Phase II: Event Free Survival and Overall Survival
Description: Event free survival is defined as the time from start of treatment to disease progression or death from any cause. Overall survival (OS) is defined as the time from start of treatment to death from any cause. A response-evaluable subject will be considered anyone who completes at least 2 cycles of therapy with documented response or documented progression of disease after at least one complete cycle of therapy but, prior to 2 complete cycles of therapy.
  A response-evaluable subject will be considered anyone who completes at least 2 cycles of therapy with documented response or documented progression of disease after at least one complete cycle of therapy but, prior to 2 complete cycles of therapy. A non-evaluable subject will be one who receives less than one complete cycle of therapy (ie. 4 infusions of ofatumumab and 21 days of lenalidomide). A non-evaluable subject will also be one that has no documented response prior to treatment withdrawal.
Time Frame: 2 years from start of treatment
Population: Six patients in Phase 1 were treated at the MTD and 34 patients enrolled in Phase II were eligible for evaluation. Data was analyzed for all patients treated at the MTD (n=40).
Measure: Number; unit: percent of participants
Groups:
- Phase II: Lemalidomide at MTD and Ofatumumab: Event free and overall survival probabilities will be computed on all patients receiving the MTD dose, including those patients in the phase I portion of the study.
Arm/Group | Phase II: Lemalidomide at MTD and Ofatumumab
Number analyzed (Participants) | 40
percent of participants
  Estimated 1 year Event Free Survival | 38
  Estimated 1 year Overall Survival | 53
  Estimated 2 year Event Free Survival | 20
  Estimated 2 year Overall Survival | 44

ADVERSE EVENTS:
Time Frame: 6 years
Groups:
- Phase I: Cohort -1: Lenalidomide: 10 mg per day.
- Phase 1: Cohort #1: Lenalidomide: 15mg per day.
- Phase 1: Cohort #2: Lenalidomide: 20mg per day.
- Phase 1: Cohort #3: Lenalidomide: 25 mg per day.
- Phase 1 & II: Event Free & Overall Survival: Event free & Overall Survival on Lenalidomide at maximum tolerated dose (MTD).
Arm/Group | Phase I: Cohort -1 | Phase 1: Cohort #1 | Phase 1: Cohort #2 | Phase 1: Cohort #3 | Phase 1 & II: Event Free & Overall Survival
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/4 | 0/0 | 0/0 | 6/36
Serious Adverse Events (participants affected / at risk) | 4/6 | 3/4 | 0/0 | 0/0 | 14/36
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 0/0 | 0/0 | 18/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Cohort -1 (N=6) | Phase 1: Cohort #1 (N=4) | Phase 1: Cohort #2 (N=0) | Phase 1: Cohort #3 (N=0) | Phase 1 & II: Event Free & Overall Survival (N=36)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Pneumonia
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and prcedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — spinal cord compression
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — deep vein thrombosis left upper extremity
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 2 (3)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — multidrug resistant pseudomonas aeurignosa
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — chronic sino-pulmonary infection
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — neutropenia
Respiratory, thoracic and medicastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Shortness of breath
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) — Neutropenia
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
confusion (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Nervous system disorders - )ther, specify (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — dysmetria
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — acute hypoxic respiratory failure
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — lactic acidosis
sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — bowel perforation
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — malignant pleural effusion
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — line infection
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — thrombocytopenia
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — positive cultures from bronch organisms; bronchoalveolar lavage positive for aspergillum in addition to candidiases
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — harsh cough
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — E. Coli bacteremia
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — acute metabolic encephalopathy, likely secondary to bacteremia
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Acute renal failure
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weakness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiatory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — reactive airway disease
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Cohort -1 (N=6) | Phase 1: Cohort #1 (N=4) | Phase 1: Cohort #2 (N=0) | Phase 1: Cohort #3 (N=0) | Phase 1 & II: Event Free & Overall Survival (N=36)
Neutrophil count decreased (Investigations) | 3 (22) | 4 (20) | 0 (0) | 0 (0) | 16 (45) — Neutropenia
Platelet count decreased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) — thrombocytopenia
White blood cell decreased (Investigations) | 1 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — leukopenia
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Investigations - Other, specify (Investigations) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — creatinine
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No